CLINICAL TRIAL: NCT05732298
Title: Theta Burst Stimulation in Pharmacologically Untreated Patients as Sole Antidepressant
Brief Title: Theta Burst Stimulation in Pharmacologically Untreated Patients as Sole Antidepressant Treatment
Acronym: TRUST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Prof. Dr., University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-3053-101
Record Dates: First submitted 2023-02-07; First posted 2023-02-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active treatment (Experimental): intermittent theta burst stimulation
  Interventions: Device: intermittend theta burst stimulation (iTBS)
- waiting list (No Intervention): patients waiting for intervention

INTERVENTIONS:
Device: intermittend theta burst stimulation (iTBS) — 600 pulses of iTBS per day with 120% resting motor threshold applied four weeks at Monday-Friday
  Other Names: repetitive transcranial magnetic stimulation
  Arms: active treatment

SUMMARY:
This is a randomized, controlled trial in which 72 patients with depressive disorder were treated in two study arms using the non-invasive brain stimulation method of intermittent thetaburst intermittent theta burst stimulation (iTBS).

This is a wait-list control study, and the arms differ in the start of the four-week treatment (either promptly i.e., at the beginning of the next week of work) or delayed (start of treatment in four weeks).

The patients to be treated are those who refuse treatment with antidepressant medications.

The effectiveness of the four-week iTBS treatment is to be evaluated in comparison to a "watchful waiting" after 4 weeks.

A interim analysis is planned after 36 patients.

ELIGIBILITY:
Inclusion Criteria:

* uni- or bipolar depression according to ICD-10
* present episode at least four weeks
* 18-70 years old
* no intake and rejection of anti-depressant medication and
* no adequate anti-depressant medication in the present episode
* no or stable non-drug anti-depressant treatment (e.g. psychotherapy)
* residency in Germany, German speaking

Exclusion Criteria:

* contraindications for transcranial magnetic stimulation (electric devices or metal parts in the body such as pacemaker
* relevant neurological or internistic diseases according to study investigator
* participation in other trials during treatment
* pregnancy or breatfeeding
* legal care and placement in a psychiatric hospital
* active suicidality

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 8 weeks
  Hamilton Depression Rating Scale (range: 0-65; higher values = worse outcome)

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | 20 weeks
  Hamilton Depression Rating Scale (range: 0-65; higher values = worse outcome)
Major Depression Inventory | 20 weeks
  Major Depression Inventory (range: 0-50; higher values = worse outcome)
World Health Organisation quality of life bref | 20 weeks
  World Health Organisation quality of life bref (range: 4-20; lower values = worse outcome)
State Trait Anxiety Inventory | 20 weeks
  State Trait Anxiety Inventory (range: 20-80 for both trait and state anxiety (two scales); higher values = worse outcome)
clinical global impression | 20 weeks
  clinical global impression (range: 0-7; higher values = worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, Prof., Principal Investigator — University Hospital of Regensburg, Department of Psychiatry and Psychotherapy at the Bezirksklinikum
Locations (1):
- Department of Psychiatry and Psychotherapy, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No